CLINICAL TRIAL: NCT00583388
Title: The Efficacy of L-arginine in Preventing Early Morning Endothelial Dysfunction
Brief Title: The Role of L-arginine in the Endothelial Dysfunction
Status: Withdrawn | Type: Observational
Why Stopped: PI is leaving the Institution, IRB will close the protocol.
Sponsor: Mayo Clinic (Other)
Responsible Party: Fatima Helena Sert Kuniyoshi, PhD (PI), Mayo Clinic
Other Study IDs: 06-008907
Record Dates: First submitted 2007-12-20; First posted 2007-12-31 (Estimated); Last update posted 2015-04-28 (Estimated); Status verified 2015-04

CONDITIONS: Healthy
Keywords: cardiology; preventive medicine; cardiovascular physiology; healthy subjects
MeSH Terms: interventions — Arginine; Ultrasonography

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — whole blood
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- A: 42 healthy subjects aged 18 to 60 will be be randomly assigned to 6 different treatment sequences.
  Interventions: Dietary Supplement: L-arginine; Device: Ultrasound

INTERVENTIONS:
Dietary Supplement: L-arginine — Each subject will be exposed to three treatments, a) 5 g of L-arginine, b) 15 g of L-arginine, and c) placebo, the sequences will be randomly assigned to the 42 volunteers. The washout period between interventions will be from one to two days.L-arginine will be mixed in 60 cc of dextrose-based syrup to blind the taste and color of the L-arginine powder.
Device: Ultrasound — Ultrasound from the brachial artery will be done on 3 occasions: at 9 pm after 4hs of fasting, at 6 am and at 11 am. The brachial artery images will be acquired above the antecubital fossa in the longitudinal plane of the artery with an ultrasound machine using a 6-MHz linear transducer. Flow-mediated vasodilatation will be assessed by the reactive hyperemia method (inflation of a blood pressure cuff around the forearm to 200 mmHg for 5 minutes and then released). The diameter of the brachial artery will be assessed 60 to 90 s after deflation of the cuff. After a 10min period a second baseline image of the brachial artery will be obtained. Non-low-mediated vasodilatation will be measured by an administration of a sublingual dose of nitroglycerin (0.4 mg).

SUMMARY:
Acute cardiac and vascular events, like heart attack and sudden cardiac death manifest a clear surge in the early morning hours around the time of waking, so that their peak onset is between 6AM and 11AM. The mechanisms are not fully understood, but we had shown that healthy subjects have impaired vascular reactivity in the early morning (endothelial dysfunction). This is associated with a decrease in nitric oxide levels (a substance that promotes vasodilatation). We also have described that vessel reactivity and the levels of this substance can recover by noon only when people breakfast.

L-arginine is a semi-essential amino acid found in large quantities in chicken, in fish, and beans and is the substrate for the production of nitric oxide Therefore we want to test if there is a beneficial effect of administration of L-arginine on the circadian pattern of vessel reactivity. Our goal is to understand why cardiovascular events are more likely to happen in the early morning and how to prevent.

The research will help us to understand the efficacy, acute effects and tolerability of high doses of L-arginine. This can lead to future research to assess long term effects of L-arginine supplements to prevent cardiovascular events in the early morning hours.

DETAILED DESCRIPTION:
Acute cardiac and vascular events, including sudden cardiac death, myocardial infarction, and stroke manifest a clear surge in the early morning hours around the time of waking, so that their peak onset is between 6 AM and 11AM. The mechanisms for this morning increase in acute cardiovascular events are not fully understood. Factors such as arousal from sleep, increased sympathetic drive, increased vasoconstrictor sensitivity and impaired endothelial function have been implicated.

We recently described the occurrence of early morning endothelial dysfunction, with blunted flow-mediated arterial dilatation in the early hours after waking. Our preliminary data suggest that this early morning endothelial dysfunction is likely due to an increased plasma levels of L-arginine endogenous inhibitor, ADMA and reducted plasma L-arginine levels, with consequent reduced availability of NO in the morning. The early morning fall in NOx levels can be potentiated by fasting and attenuated by a low-nitrate, protein rich breakfast. Because the production of NO depends in part on the availability of L-arginine, methods to maintain an adequate level of plasma L-arginine in the early morning are needed. We propose to assess the efficacy of high doses of L-arginine in preventing early morning endothelial dysfunction.

The primary aim is to examine the effects of high doses of L-arginine on morning changes in nitric oxide and endothelial function. Our hypotheses are:

1. That L-arginine administered orally prior to sleep will prevent the early morning decline in plasma levels of L-arginine and nitric oxide; 2. That L-arginine administered prior to sleep will attenuate or prevent the early morning decline in endothelial function; and 3. That the effects of L-arginine, taken prior to sleep, on plasma levels of L-arginine and nitric oxide and on endothelial function will be more marked with 15 grams of L-arginine versus 5 grams of L-arginine or placebo, indicative of a dose response effect.

Our secondary aim is to identify the short-term tolerability and safety of two different doses of L-arginine. Our hypothesis is that subjects taking high doses of L-arginine (15 grams) will not have significant symptoms or adverse changes in vital signs.

ELIGIBILITY:
Inclusion Criteria:

* healthy subjects

Exclusion Criteria:

* renal disease; liver disease, sleep disorders, smokers, using chronic medications

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: community sample
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2010-06; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Virend K Somers, MD, PhD, Study Chair — Mayo Clinic